CLINICAL TRIAL: NCT06463041
Title: Effects of Low-intensity Office Training and Standing Work on Health and Functional Performances Among Female Computer Users: A Randomized Controlled Trial
Brief Title: How Does Implementing a GetUp Assist Device in Addition to a Daily Low-intensity Functional or Traditional Training Program Affect Norwegian Female Office Workers' Physical Health After 12 Weeks?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Lasse Engberg Treu Lassen, Ph.D., Aalborg University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 438957
Record Dates: First submitted 2024-06-08; First posted 2024-06-17 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Neck, Shoulder and Arm Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Functional training group (Experimental): Functional training group that will perform a short, low-intensity, 10-minute hole-body exercise program per day before the lunch break, in addition to following the getup assistance during the working day.
  Interventions: Other: Experimental, comparator and control
- Traditional training group (Active Comparator): Traditional training group that will perform a short, low-intensity, 10-minute hole-body exercise program per day before the lunch break, in addition to following the getup assistance during the working day.
  Interventions: Other: Experimental, comparator and control
- Negative control (No Intervention): Control group. A group that is not treated.

INTERVENTIONS:
Other: Experimental, comparator and control — How does implementing a GetUp Assist device in addition to a daily low-intensity functional or traditional training program affect Norwegian female office workers' physical health after 12 weeks?
  Arms: Functional training group; Traditional training group

SUMMARY:
This study aims to quantify the effect of daily transition routines between sitting and standing behaviour with an additional daily low-intensity traditional or functional training program on the physical health of sedentary Norwegian female workers after 12 weeks of implementation into their working environment.

ELIGIBILITY:
Inclusion Criteria:

* Females are included in this study due to the approximately twice-high prevalence of work-related musculoskeletal disorders.
* No experience with office fit training or participation in an ongoing similar training intervention is allowed.
* Working more than 6 hours a day at a computer workstation
* Physical inactivity (less than two sessions or bouts of exercise totalling 30 minutes/week).
* Musculoskeletal complaints are accepted as long as the pain is not a restricting factor. when performing the testing and training intervention exercises.

Exclusion Criteria:

* Participants not able to perform the testing battery.

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 58 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2024-12-22 (Actual); Study Completion 2024-12-22 (Actual)

PRIMARY OUTCOMES:
Norwegian Short-Form Health Survey (SF-36) | 3 months
  Measure (i) physical function, (ii) Energy/fatigue, (iii) pain, and (iv) general health
Neck and shoulder trouble questionnaire from the Nordic musculoskeletal questionnaire | 3 months
  Measure neck-shoulder discomfort
Numeric rating scale | 3 months
  Measure neck-shoulder discomfort from 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable
Y-balance test | 3 months
  Quantify dynamic postural control
The Danish step test | 3 months
  Estimating cardiorespiratory fitness
Chair-sit-and-reach test | 3 months
  Measuring hamstrings flexibility
Back scratch test | 3 months
  Measuring upper-body/ shoulder flexibility
CS-30 test | 3 months
  Measuring lower-body strength
Hand Grip Strength test | 3 months
  Measuring hand Grip Strength

CONTACTS AND LOCATIONS:
Locations (1):
- SSA Steinkjer, Steinkjer, Nord-Trøndelag, Norway